CLINICAL TRIAL: NCT05239156
Title: Open, Non-comparative, Multicentre Clinical Investigation to Evaluate the Performance and Safety of the Medical Device Janesse® (Hyaluronic Acid-dermal Filler) in the Treatment of Facial Dermal Tissue Defects
Brief Title: Evaluating the Performance and Safety of the Medical Device Janesse in the Treatment of Facial Dermal Tissue Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPIRA/0221/MD
Record Dates: First submitted 2022-01-17; First posted 2022-02-14 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-03

CONDITIONS: Cicatrix; Lipodystrophy; Plaque
MeSH Terms: conditions — Cicatrix; Lipodystrophy; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, non-randomized clinical investigation
Masking Description: Sixteen patients will be administered Janesse® 15 (Cross-linked Hyaluronic Acid) for the treatment of minor facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects).
  Sixteen patients will be administered Janesse® 20 (Cross-linked Hyaluronic Acid) for the treatment of medium-sized facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects).
  Sixteen patients will be administered Janesse® 25 (Cross-linked Hyaluronic Acid) for the treatment of major facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Janesse 15 (Experimental): Sixteen patients will be administered Janesse® 15 (Cross-linked Hyaluronic Acid) for the treatment of minor facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects).
  Interventions: Device: Janesse
- Janesse 20 (Experimental): Sixteen patients will be administered Janesse® 20 (Cross-linked Hyaluronic Acid) for the treatment of medium-sized facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects).
  Interventions: Device: Janesse
- Janesse 25 (Experimental): Sixteen patients will be administered Janesse® 25 (Cross-linked Hyaluronic Acid) for the treatment of major facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects).
  Interventions: Device: Janesse

INTERVENTIONS:
Device: Janesse — Device: Janesse® is a sterile, injectable, non-pyrogenic, re-absorbable medical product made of reticulated hyaluronic acid of non-animal origin, produced via bacterial fermentation.
  The subjects will receive at baseline the first investigational medical device by the Investigator in accordance with the clinical investigation plan.

SUMMARY:
The Research Question of the present study is the following: in a population of men and women presenting facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects) will cross-linked hyaluronic acid (Janesse®) significantly decrease and / or improve the appearance of these defects, results observed after 4, 8 and 12 weeks?

DETAILED DESCRIPTION:
Janesse® action is to increase the volume of dermal-epidermal tissue, based on the natural ability of hydrophilic hyaluronic acid molecules to bind to an amount of water many times greater than their weight. This allows to fill the intradermal spaces and integrate the intercellular matrix, conferring turgidity to the tissues. The cross-linking of the hyaluronic acid contained in the product has the effect of more stable and durable filling over time. These characteristics allow Janesse® to be used as a temporary filler for subcutaneous areas to correct small defects in the dermal tissue due to lipodystrophies or the presence of fibrotic tissues as scars, caused by pathologies or trauma.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with age ≥ 18 and ≤ 65 years.
2. Patients with facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects) caused both by pathologies or trauma, seeking tissue augmentation treatment and willing to receive Hyaluronic Acid Filler.
3. Patients who agree to discontinue any other dermatological treatment and procedures during the study.
4. Patients willing to provide signed informed consent to clinical investigation participation.
5. Patients able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

1. Past or current bleeding disorders.
2. Use of aspirin and antiplatelet agents a week prior to treatment.
3. Prior or planned use of topical injection to the face (steroid, retinoid: applicable only to drugs, not applicable to cosmetics), within 4 weeks prior to screening or during this study (steroid ointment for therapeutic objectives is allowed for short -term use of ≤14 consecutive days.).
4. Use of immunosuppressive, chemotherapies, or systemic corticosteroids within 12 weeks from screening.
5. History of anaphylaxis or severe complicated allergy symptoms.
6. Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders or previous mental disorders that may significantly affect the study.
7. Known hypersensitivity skin reaction to hyaluronic acid or hypersensitivity skin reaction to the investigational device based on intradermal test results at visit 1.
8. Evidence or history of autoimmune disease or compromised immune system.
9. Treatment with anticoagulants, thrombolytics, or platelet inhibitors within 1 week prior to study participation.
10. Prior permanent fillers or fat graft procedures around facial dermal tissue defects.
11. Facial dermal tissue defects correction procedures (e.g., botulinum toxin A injection, face lift, soft tissue augmentation, medium-depth peel, dermal photo-rejuvenation, etc.) around infraorbital region within 6 months prior to study participation.
12. History of hypersensitivity to local anaesthetic of amide type or HA.
13. History of keloid formation or hypertrophic scar on the face.
14. Evidence of active infection on the face.
15. Wound, skin disorder or infection around facial dermal tissue defects that may affect the efficacy assessment.
16. Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study. *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
17. Need to exposure to the sun, UV rays and extreme conditions of heat for at least a week after the treatment.
18. Need to have direct or indirect contact with quaternary ammonium salts during the study.
19. As with all dermal filler procedures, the product should not be used in vascular rich areas. Using the product at sites such as Glabella and nose may inadvertently be injected into the blood vessels, resulting in symptom of vessel occlusion such as colour vision deficiency and blindness.
20. Patients with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the study.
21. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
POSAS score assessed by Investigator and patient | 8 weeks
  To evaluate the overall performance of the medical dermal filler Janesse® in treating facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects) in terms of change in Patient and Observer Scar Assessment Scale (POSAS) score [Draaijers, 2004; van de Kar, 2005], assessed by Investigators and patients at 8 weeks (56 days) after the initiation of treatment, compared to Visit 1 (day 0).
POSAS score assessed by Investigator and patient | 4 weeks
  To evaluate the overall performance of the medical dermal filler Janesse® in treating facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects) in terms of change in Patient and Observer Scar Assessment Scale (POSAS) score [Draaijers, 2004; van de Kar, 2005], assessed by Investigators and patients at 4 weeks (28 days) after the initiation of treatment, compared to Visit 1 (day 0).
POSAS score assessed by Investigator and patient | 12 weeks
  To evaluate the overall performance of the medical dermal filler Janesse® in treating facial dermal tissue defects (scars, depressed plaques, and lipodystrophy defects) in terms of change in Patient and Observer Scar Assessment Scale (POSAS) score [Draaijers, 2004; van de Kar, 2005], assessed by Investigators and patients at 12 weeks (84 days) after the initiation of treatment, compared to Visit 1 (day 0).
Investigator Global Assessment of Performance (IGAP) | 12 weeks
  To evaluate the global performance of product assessed by Investigator through photos taken at each visit (IGAP), at week 12 (day 84), compared to Visit 1 (day 0).
Adverse Event incidence | 12 weeks
  To evaluate the safety of the device trough Adverse Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Serious Adverse Event incidence | 12 weeks
  To evaluate the safety of the device trough Serious Adverse Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Adverse Device Event incidence | 12 weeks
  To evaluate the safety of the device trough Adverse device event incidence assessed by Investigators at all visits and reported according to the current legislation.
Serious Adverse Device Event incidence | 12 weeks
  To evaluate the safety of the device trough Serious Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation.

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale evaluated by the patient (GAIS) | 12 weeks
  To evaluate general appearance after treatment assessed by the patient at 4, 8 and 12 weeks (28, 56 and 84 days) using the Global Aesthetic Improvement Scale (GAIS) [Kim, 2016], [Kopera, 2015 - 2018], [McCall-Perez, 2011], [Savoia, 2015]. The scale evaluates the appearance from 1 (very much improved) to 5 (worse than original condition) .
Treatment satisfaction assessment by the patient | 12 weeks
  To assess the patient satisfaction at 4, 8 and 12 weeks (28, 56 and 84 days), providing their degree of satisfaction with the treatment on a four-point scale (very satisfied, satisfied, moderately satisfied, or not satisfied)
Investigator Global Assessment of Safety (IGAS) | 12 weeks
  To evaluate the global safety of product assessed by Investigator (IGAS), at week 12 (day 84), compared to Visit 1 (day 0), providing the safety on a four point scale from 4 meaning poor safety to 1 meaning very good safety.
Patient Global Assessment of Safety (PGAS) | 12 weeks
  To evaluate the global safety of product assessed by the patient (PGAS), at week 12 (day 84), compared to Visit 1 (day 0), providing the safety on a four point scale from 4 meaning poor safety to 1 meaning very good safety.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Fratila, Principal Investigator — SCM Dr. Rosu
Locations (1):
- SCM Dr. Rosu, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Eming SA, Martin P, Tomic-Canic M. Wound repair and regeneration: mechanisms, signaling, and translation. Sci Transl Med. 2014 Dec 3;6(265):265sr6. doi: 10.1126/scitranslmed.3009337. PMID 25473038
- [Background] Almeida A, Sampaio G. Hyaluronic acid in the rejuvenation of the upper third of the face: review and update - Part 1. 2018.
- [Background] Ascher B, Bayerl C, Brun P, Kestemont P, Rzany B, Poncet M, Guennoun M, Podda M. Efficacy and safety of a new hyaluronic acid dermal filler in the treatment of severe nasolabial lines - 6-month interim results of a randomized, evaluator-blinded, intra-individual comparison study. J Cosmet Dermatol. 2011 Jun;10(2):94-8. doi: 10.1111/j.1473-2165.2011.00550.x. PMID 21649813
- [Background] Barnes LA, Marshall CD, Leavitt T, Hu MS, Moore AL, Gonzalez JG, Longaker MT, Gurtner GC. Mechanical Forces in Cutaneous Wound Healing: Emerging Therapies to Minimize Scar Formation. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):47-56. doi: 10.1089/wound.2016.0709. PMID 29392093
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Brandt FS, Cazzaniga A. Hyaluronic acid gel fillers in the management of facial aging. Clin Interv Aging. 2008;3(1):153-9. doi: 10.2147/cia.s2135. PMID 18488885
- [Background] Bukhari SNA, Roswandi NL, Waqas M, Habib H, Hussain F, Khan S, Sohail M, Ramli NA, Thu HE, Hussain Z. Hyaluronic acid, a promising skin rejuvenating biomedicine: A review of recent updates and pre-clinical and clinical investigations on cosmetic and nutricosmetic effects. Int J Biol Macromol. 2018 Dec;120(Pt B):1682-1695. doi: 10.1016/j.ijbiomac.2018.09.188. Epub 2018 Oct 1. PMID 30287361
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448
- [Background] Rippa AL, Kalabusheva EP, Vorotelyak EA. Regeneration of Dermis: Scarring and Cells Involved. Cells. 2019 Jun 18;8(6):607. doi: 10.3390/cells8060607. PMID 31216669
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] De Boulle K, Heydenrych I. Patient factors influencing dermal filler complications: prevention, assessment, and treatment. Clin Cosmet Investig Dermatol. 2015 Apr 15;8:205-14. doi: 10.2147/CCID.S80446. eCollection 2015. PMID 25926750
- [Background] Dong J, Gantz M, Goldenberg G. Efficacy and safety of new dermal fillers. Cutis. 2016 Nov;98(5):309-313. PMID 28040813
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628
- [Background] Fitzgerald R, Graivier MH, Kane M, Lorenc ZP, Vleggaar D, Werschler WP, Kenkel JM. Update on facial aging. Aesthet Surg J. 2010 Jul-Aug;30 Suppl:11S-24S. doi: 10.1177/1090820X10378696. PMID 20844296
- [Background] Freedberg et al. Fitzpatrick's Dermatology In General Medicine (Two Vol. Set) 6th edition (May 23, 2003
- [Background] Funt D, Pavicic T. Dermal fillers in aesthetics: an overview of adverse events and treatment approaches. Plast Surg Nurs. 2015 Jan-Mar;35(1):13-32. doi: 10.1097/PSN.0000000000000087. PMID 25730536
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Gottfried Lemperle, M.D., Ph.D., Ralph E. Holmes, M.D., Steven R. Cohen, M.D., and Stefan M. Lemperle, M.D., A Classification of Facial Wrinkles, Division of Plastic Surgery, University of California, and FACESplus, Inc. Received for publication September 15, 2000; revised January 5, 2001.
- [Background] Grablowitz D, Ivezic-Schoenfeld Z, Federspiel IG, Gehl B, Kopera D, Prinz M. Long-term effectiveness of a hyaluronic acid soft tissue filler in patients with facial lipoatrophy, morphological asymmetry, or debilitating scars. J Cosmet Dermatol. 2020 Oct;19(10):2536-2541. doi: 10.1111/jocd.13454. Epub 2020 Jun 22. PMID 32333705
- [Background] Jiang LI, Stephens TJ, Goodman R. SWIRL, a clinically validated, objective, and quantitative method for facial wrinkle assessment. Skin Res Technol. 2013 Nov;19(4):492-8. doi: 10.1111/srt.12073. Epub 2013 Jun 10. PMID 23750828
- [Background] Kim BW, Moon IJ, Yun WJ, Chung BY, Kim SD, Lee GY, Chang SE. A Randomized, Evaluator-Blinded, Split-Face Comparison Study of the Efficacy and Safety of a Novel Mannitol Containing Monophasic Hyaluronic Acid Dermal Filler for the Treatment of Moderate to Severe Nasolabial Folds. Ann Dermatol. 2016 Jun;28(3):297-303. doi: 10.5021/ad.2016.28.3.297. Epub 2016 May 25. PMID 27274627
- [Background] Kopera D, Ivezic-Schoenfeld Z, Federspiel IG, Grablowitz D, Gehl B, Prinz M. Treatment of facial lipoatrophy, morphological asymmetry, or debilitating scars with the hyaluronic acid dermal filler Princess(R) FILLER. Clin Cosmet Investig Dermatol. 2018 Nov 27;11:621-628. doi: 10.2147/CCID.S181964. eCollection 2018. PMID 30568476
- [Background] Kopera D, Palatin M, Bartsch R, Bartsch K, O'Rourke M, Holler S, Baumgartner RR, Prinz M. An open-label uncontrolled, multicenter study for the evaluation of the efficacy and safety of the dermal filler Princess VOLUME in the treatment of nasolabial folds. Biomed Res Int. 2015;2015:195328. doi: 10.1155/2015/195328. Epub 2015 Mar 3. PMID 25821787
- [Background] Kuhne U, Esmann J, von Heimburg D, Imhof M, Weissenberger P, Sattler G. Safety and performance of cohesive polydensified matrix hyaluronic acid fillers with lidocaine in the clinical setting - an open-label, multicenter study. Clin Cosmet Investig Dermatol. 2016 Oct 20;9:373-381. doi: 10.2147/CCID.S115256. eCollection 2016. PMID 27799807
- [Background] Lorenc ZP, Bank D, Kane M, Lin X, Smith S. Validation of a four-point photographic scale for the assessment of midface volume loss and/or contour deficiency. Plast Reconstr Surg. 2012 Dec;130(6):1330-1336. doi: 10.1097/PRS.0b013e31826d9fa6. PMID 23190816
- [Background] Mashiko T, Kinoshita K, Kanayama K, Feng J, Yoshimura K. Perpendicular Strut Injection of Hyaluronic Acid Filler for Deep Wrinkles. Plast Reconstr Surg Glob Open. 2015 Dec 9;3(11):e567. doi: 10.1097/GOX.0000000000000552. eCollection 2015 Nov. PMID 26893992
- [Background] McCall-Perez F, Stephens TJ, Herndon JH Jr. Efficacy and tolerability of a facial serum for fine lines, wrinkles, and photodamaged skin. J Clin Aesthet Dermatol. 2011 Jul;4(7):51-4. PMID 21779421
- [Background] Rivkin AZ. Volume correction in the aging hand: role of dermal fillers. Clin Cosmet Investig Dermatol. 2016 Aug 30;9:225-32. doi: 10.2147/CCID.S92853. eCollection 2016. PMID 27621659
- [Background] Rumsey N. Psychosocial adjustment to skin conditions resulting in visible difference (disfigurement): What do we know? Why don't we know more? How shall we move forward? Int J Womens Dermatol. 2017 Dec 15;4(1):2-7. doi: 10.1016/j.ijwd.2017.09.005. eCollection 2018 Mar. PMID 29872669
- [Background] Rzany B, Cartier H, Kestemont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC, Ma YM. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol Surg. 2012 Jul;38(7 Pt 2):1153-61. doi: 10.1111/j.1524-4725.2012.02470.x. PMID 22759252
- [Background] Savoia A., Onori N., Bladi A., Efficacy of Skinfill plus filler in the management of facial aging: a multicenter, post-marketing clinical study, Biomedical Dermatology volume 2, Article number: 2 (2018).
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135
- [Background] Sudha PN, Rose MH. Beneficial effects of hyaluronic acid. Adv Food Nutr Res. 2014;72:137-176. doi: 10.1016/B978-0-12-800269-8.00009-9. PMID 25081082
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Van Dyke S, Hays GP, Caglia AE, Caglia M. Severe Acute Local Reactions to a Hyaluronic Acid-derived Dermal Filler. J Clin Aesthet Dermatol. 2010 May;3(5):32-5. PMID 20725567